CLINICAL TRIAL: NCT00334451
Title: Remote Active Monitoring in Patients With Heart Failure
Brief Title: RAPID-RF: Remote Active Monitoring in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-CA-030206-H; RAPID RF
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Remote Monitoring; Implantable Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The RAPID-RF Registry aims to characterize LATITUDE® Patient Management's alert feature: LATITUDE Active Monitoring™ by evaluating type and frequency of alert notifications and alert-related medical interventions. This registry will also assess clinical outcomes including quality of life and New York Heart Association Class changes over time, mortality, hospitalizations and heart failure-related event rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for a Guidant RF-enabled CRT-D device (e.g. CONTAK RENEWAL 3 RF family of CRT-D devices) which is compatible with the LATITUDE Communicator. Indications include: NYHA Class III, IV; EF of ≤ 35%; QRS duration of ≥ 120 ms; and optimized pharmacologic therapy
* Patients who have an analog telephone line compatible with the LATITUDE Communicator. The LATITUDE Communicator must be placed within 8 feet of where they sleep for successful remote interrogations to occur.
* Patients who receive the study components including the LATITUDE Communicator, weight scale, and blood pressure monitor
* Patients who are willing and capable of providing informed consent prior to implant and willing to participate in the RAPID-RF Registry
* Patients who remain in the clinical care of a RAPID-RF investigator at approved centers

Exclusion Criteria:

* Patients who are expected to receive a heart transplant during the course of the study
* Patients who have received or who will receive a tricuspid valve prosthesis during the course of the study
* Patients who have previously received an implantable cardiac resynchronization device (e.g., biventricular pacemaker or biventricular ICD)
* Patients whose life expectancy is less than 12 months
* Patients who are currently enrolled in another observational registry or investigational study that could directly impact the treatment or outcome of the RAPID-RF Registry. Contact Guidant's Clinical Application Research Study (CARS) department to determine eligibility.
* Patients who are younger than 18 years of age
* Patients who are pregnant or plan to become pregnant during the study
* Patients who are unable or refuse to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics, heart failure clinics, hospitals
Sampling Method: Non-Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Saxon, MD, Principal Investigator — University of Southern California; John P Boehmer, MD, Principal Investigator — Hershey Medical Center, Hershey, PA
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

REFERENCES:
- [Derived] Saxon LA, Boehmer JP, Neuman S, Mullin CM. Remote Active Monitoring in Patients with Heart Failure (RAPID-RF): design and rationale. J Card Fail. 2007 May;13(4):241-6. doi: 10.1016/j.cardfail.2006.12.004. PMID 17517341